CLINICAL TRIAL: NCT06509711
Title: Comparative Effects Of Mud Based Plyometric Jump Training With And Without High Intensity Interval Training on Speed, Power and Calf Girth of Volleyball Players
Brief Title: Comparative Effects Of Mud Based Plyometric Jump Training on Volleyball Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR &AHS/23/0475
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Sports Physical Therapy
Keywords: calf girth; mud-based Plyometric training; speed

STUDY DESIGN:
Intervention Model Description: randomized clinical trials
Who Masked: Outcomes Assessor
Masking Description: single (outcome assessor) who take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLYOMETRICS jump training with HIIT (Experimental): Alternate Jump Lunge (4 REPS, 3 SETS with 25 SECONDS recovery period between each SET )
  Split squat jump (4 REPS, 3 SETS with 25 SECONDS recovery between each SET) Pop Squat (4 REPS, 3 SETS with 25 SECONDS recovery period between each set)
  Interventions: Other: PLYOMETRICS jump training with HIIT (4 weeks,3 sessions per week)
- PLYOMETRICS JUMP TRAINING WITHOUT HIIT (Experimental): Plate pogo (4 reps, 3 sets) Broad jump( 4reps,3 sets)
  Interventions: Other: PLYOMETRICS JUMP TRAINING WITHOUT HIIT (4weeks, 3sessions Per week)

INTERVENTIONS:
Other: PLYOMETRICS jump training with HIIT (4 weeks,3 sessions per week) — First set of drills 6 x 40-cm hurdle jumps +5-s sprint* at 130% of aerobic maximum speed. Second set of drills 6 x 30-cm hurdle jumps with extended legs + 5-s sprint at 130% of aerobic maximum speed. Third set of drills 6 x horizontal jumps + 5-s sprint at 130% of aerobic maximum speed. Fourth set of drills 3 right-leg and 3left-leg hops +5-s sprint at 130% of aerobic maximum speed. Each drills set was performed 2 times in a row. Afterwards, 10 seconds of rest were allowed. Thereafter, this sequence of effort-rest was repeated 8 times. After then, a 3-5 min recovery period was allowed before commencing the next drills set;
  Arms: PLYOMETRICS jump training with HIIT
Other: PLYOMETRICS JUMP TRAINING WITHOUT HIIT (4weeks, 3sessions Per week) — Plate pogo (4 reps, 3 sets) Broad jump( 4reps,3 sets)
  Arms: PLYOMETRICS JUMP TRAINING WITHOUT HIIT

SUMMARY:
Volleyball is a high-intensity, anaerobic sport that alternates between brief rest intervals and explosive movements in both vertical and horizontal planes. Therefore, it is believed that essential components of successful athletic performance are explosive strength, speed and power which are defined as the neuro- muscular system of an individual's ability to manifests training the shortest amount of time. The complex movement of a vertical jump necessitates the coordination of multiple muscles in the arms, legs, and trunk. Being aware that a five-set volleyball match requires more than 250 jumps from each player. Eight weeks of plyometric jump training on mud and other unstable surfaces caused some changes in the biomechanical variables and physical fitness related to volley ball performance in volley ball players. Thus, by adding more high-intensity training, elite volleyball players can maximize their physical performance level during the competitive season.

DETAILED DESCRIPTION:
This study was randomized clinical trial and was conducted in Pakistan Sports Board in duration of 10 months. Non-probability convenient sampling technique was used. Sample size was 30 calculated by G-power using 50-m sprint as variable. Participants were recruited into 2 equal groups by the process of randomization according to inclusion and exclusion criteria. One group performed mud based plyometric jump training with high intensity interval training which included alternate jump lunge, split squat jump and pop squat jump 4 repetitions, 3 sets and other performed mud based plyometric jump training without high intensity interval training which included plate pogo and broad jump 4 REPS, 3 SETS. Data was analyzed by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Age:17-35years
* Male Volleyball players
* 1 Repetition Maximum (RM) of 10kg
* BMI in the range of 18.5 to 24.9
* Players had game experience of at least 2years

Exclusion Criteria:

* Musculoskeletal issues(Jumper's knee, Foot and ankle injuries, Patellar tendinopathy, Ligamentous and meniscal injury, Bone deformity, Fractures of lower limb)
* Cardiac and Pulmonary disorder
* Vestibular and visual disorder

Ages: 17 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-09-26 (Estimated)

PRIMARY OUTCOMES:
speed | 0 week, 6 week, 12 week
  speed of athlete measure by 50-m linear sprint
calf girth | 0 week, 6 week, 12 week
  it is measured by Gulick tape
power | 0 week, 6 week, 12 week
  it is measured by vertical jump

CONTACTS AND LOCATIONS:
Overall Officials: Atif Javed, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Markovic G. Does plyometric training improve vertical jump height? A meta-analytical review. Br J Sports Med. 2007 Jun;41(6):349-55; discussion 355. doi: 10.1136/bjsm.2007.035113. Epub 2007 Mar 8. PMID 17347316
- [Background] Bobbert MF. Drop jumping as a training method for jumping ability. Sports Med. 1990 Jan;9(1):7-22. doi: 10.2165/00007256-199009010-00002. PMID 2408119
- [Background] Thomas K, French D, Hayes PR. The effect of two plyometric training techniques on muscular power and agility in youth soccer players. J Strength Cond Res. 2009 Jan;23(1):332-5. doi: 10.1519/JSC.0b013e318183a01a. PMID 19002073
- [Background] Chen L, Zhang Z, Huang Z, Yang Q, Gao C, Ji H, Sun J, Li D. Meta-Analysis of the Effects of Plyometric Training on Lower Limb Explosive Strength in Adolescent Athletes. Int J Environ Res Public Health. 2023 Jan 19;20(3):1849. doi: 10.3390/ijerph20031849. PMID 36767213
- [Background] Kons RL, Orssatto LBR, Ache-Dias J, De Pauw K, Meeusen R, Trajano GS, Dal Pupo J, Detanico D. Effects of Plyometric Training on Physical Performance: An Umbrella Review. Sports Med Open. 2023 Jan 10;9(1):4. doi: 10.1186/s40798-022-00550-8. PMID 36625965
- [Background] Silva AF, Clemente FM, Lima R, Nikolaidis PT, Rosemann T, Knechtle B. The Effect of Plyometric Training in Volleyball Players: A Systematic Review. Int J Environ Res Public Health. 2019 Aug 17;16(16):2960. doi: 10.3390/ijerph16162960. PMID 31426481
- [Background] Ahmadi M, Nobari H, Ramirez-Campillo R, Perez-Gomez J, Ribeiro ALA, Martinez-Rodriguez A. Effects of Plyometric Jump Training in Sand or Rigid Surface on Jump-Related Biomechanical Variables and Physical Fitness in Female Volleyball Players. Int J Environ Res Public Health. 2021 Dec 11;18(24):13093. doi: 10.3390/ijerph182413093. PMID 34948702
- [Background] Hoffmann JJ Jr, Reed JP, Leiting K, Chiang CY, Stone MH. Repeated sprints, high-intensity interval training, small-sided games: theory and application to field sports. Int J Sports Physiol Perform. 2014 Mar;9(2):352-7. doi: 10.1123/ijspp.2013-0189. Epub 2013 May 22. PMID 23751941